CLINICAL TRIAL: NCT06864624
Title: Sunvozertinib as Neoadjuvant and Adjuvant Therapy in Stage II-IIIB Non-small-cell Lung Cancer Patients With EGFR Exon 20 Insertion Mutation: a Single-arm, Phase 2 Study (WU-KONG20)
Brief Title: Perioperative Treatment of Sunvozertinib in Stage II-IIIB NSCLC
Acronym: WU-KONG20
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202412-18
Record Dates: First submitted 2025-01-14; First posted 2025-03-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NSCLC
Keywords: sunvozertinib; neoadjuvant; adjuvant; EGFR exon20 insertion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sunvozertinib (Experimental): Patients will receive neoadjuvant sunvozertinib for 12 weeks, and continue adjuvant sunvozertinib after surgery until disease relapse, unacceptable toxicity, or the end of 2-years adjuvant treatment.
  Interventions: Drug: Sunvozertinib

INTERVENTIONS:
Drug: Sunvozertinib — Neoadjuvant stage: 300mg for 12 weeks Adjuvant stage: 300mg for first 4 weeks, then 150mg for up to 2 years

SUMMARY:
This is a single-arm, phase 2 study to investigate the efficacy and safety of sunvozertinib as neoadjuvant and adjuvant treatment for stage II-IIIB non-small-cell lung cancer patients with EGFR exon20 insertion mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must understand the requirements and content of the clinical trial and provide a handwritten signed and dated informed consent.
2. Age ≥ 18 years old.
3. Non-small cell lung cancer confirmed by histopathology or cytology, clinical stage II, IIIA or IIIB (N2) assessed by the investigator according to AJCC 8th edition.
4. EGFR exon 20 insertion mutation confirmed by an approved local laboratory.
5. No disease progression in the past two weeks of signing the informed consent form and a score of 0-1 according to the ECOG criteria, and no significant progression within 2 weeks before the first dose.
6. At least one measurable target lesion according to RECIST v1.1.
7. Adequate bone marrow and other organ reserve:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Platelets ≥ 100 × 109/L
   * Hemoglobin ≥ 9 g/dL
   * Total bilirubin ≤ 1.5 ×ULN; in patients with Gilbert syndrome, total bilirubin ≤ 3 × ULN
   * ALT≤ 2.5 × ULN and AST≤ 2.5 × ULN
   * Creatinine ≤ 1.5 × ULN, and creatinine clearance calculated the Cockcroft-Gault method ≥ 60 mL/min
   * International normalized ratio (INR) ≤ 1.5 × ULN
   * Partial thromboplastin time (APTT) ≤ 1.5 × ULN
8. Male patients who wish to have children should use barrier contraception (such as condoms) during the clinical trial period and 6 months after the last dose. Male patients should not donate sperm during the clinical trial period and 6 months after the last dose.
9. Female patients should take contraceptive measures from the start of screening to the 6 weeks after last dose, should not breastfeed, and should have a negative pregnancy test (blood or urine β-human chorionic gonadotropin) at screening.

Exclusion Criteria:

1. Patients who have received the following treatments must be excluded:

   * Any systemic anti-tumor treatment, including radiotherapy;
   * Other drugs in the development stage, if the medication does not exceed 28 days and has not undergone any tumor assessment, the medication must be stopped for more than 5 half-lives and the patient can be enrolled after consultation with the investigator.
   * Traditional Chinese medicine and other drugs with strong P450 (CYP)3A4 inhibitory or inducing effects are currently being used or cannot be stopped. There must be a washout period of at least 1 week before the first dose.
2. A history of other malignant tumors other than lung cancer within 2 years (except for basal cell carcinoma of the skin or in situ cervical cancer that has been adequately treated and has no evidence of recurrence during the screening period).
3. Before the first dose, there are adverse events of CTCAE > 1 grade (except for any degree of alopecia) caused by previous treatment (such as diagnostic puncture, use of other drugs, etc.).
4. History of stroke or intracranial hemorrhage within 6 months before the first dose.
5. According to the investigator's judgment, the presence of any severe or poorly controlled systemic disease, including any of the following poorly controlled heart-related diseases or abnormalities:

   * The resting electrocardiogram shows a calibrated QTc interval (QTcF) > 470 msec
   * The resting electrocardiogram shows any serious abnormalities in heart rhythm, conduction or pattern, such as complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 msec
   * Any factors that can cause QTcF prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of QT syndrome or other sudden death diseases under 40 years old, or other diseases known to cause QT prolongation
   * Suffering from atrial fibrillation (except for drug-induced and recovered after discontinuation of the drug)
   * Myocardial infarction within 6 months before the first dose, New York Heart Association grade 2 congestive heart failure, or arrhythmias that are not well controlled by drugs
6. Patients with a history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid hormone treatment, or any clinically active interstitial lung disease, or immune pneumonitis caused by immunotherapy.
7. Patients with refractory nausea and vomiting, chronic gastrointestinal diseases, difficulty in swallowing medication, or previous intestinal resection that prevents adequate absorption of sunvozertinib.
8. Women who are breastfeeding or pregnant.
9. Patients who are allergic to the drug components of sunvozertinib.
10. Patients who are assessed by the investigator as being unable to undergo clinical trials, unable to tolerate surgery, or who may lack compliance with clinical trials should not participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of neoadjuvant therapy | From enrollment to the end of neoadjuvant therapy at 12 weeks
  Complete response (CR) or partial response (PR) per investigator assessment according to RECIST 1.1

SECONDARY OUTCOMES:
Major pathological response (MPR) | Pathological detection within 1month after surgery
Pathological complete response (pCR) | Pathological detection within 1 month after surgery
Downstaging rate of N2 lymph nodes | From enrollment to the end of neoadjuvant therapy at 12 weeks
Disease control rate (DCR) of neoadjuvant therapy | From enrollment to the end of neoadjuvant therapy at 12 weeks
Event free survival (EFS) | From date of enrollment until the date of first documented disease progression, relapse, or death due to any cause progression, whichever came first, assessed up to 60 months
Disease free survival (DFS) | From date of surgical resection until the date of first documented disease relapse or death due to any cause , whichever came first, assessed up to 56 months
Overall survival (OS) | From date of enrollment until the date of death due to any cause , assessed up to 84 months
Adverse events | From date of enrollment until the end of the study, assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Tangdu Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No